CLINICAL TRIAL: NCT01636479
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Biological Activity of SAR405838 in Patients With Advanced Cancer
Brief Title: Phase 1 Safety Testing of SAR405838
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED12318; 2012-000733-39; U1111-1127-2911 (Other: UTN)
Record Dates: First submitted 2012-07-02; First posted 2012-07-10 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — SAR405838

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR405838 (Experimental): SAR405838 in escalating doses
  Interventions: Drug: SAR405838

INTERVENTIONS:
Drug: SAR405838 — Pharmaceutical form: Capsule Route of administration: Oral

SUMMARY:
Primary Objectives:

* To determine safety and the maximum tolerated dose (MTD) of SAR405838 through the characterization of dose-limiting toxicities (DLTs).
* To assess biological activities in patients with dedifferentiated liposarcoma during MTD cohort expansion.

Secondary Objectives:

* Pharmacokinetic (PK) profile of SAR405838.
* Biomarkers in association with SAR405838.
* Anti-tumor activity in response to SAR405838.
* Food effect on SAR405838 PK.
* Compliance with SAR405838 treatment.
* Cytochrome P450 3A4/5 (CYP3A4/5) activity.

DETAILED DESCRIPTION:
Total duration of study participation for each patient will be one month screening followed by treatment until precluded by toxicity, noncompliance, progression, or death.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor for which no further effective standard treatment is available. Patients with lymphomas may be enrolled.
* For dose escalation, tumor type that has high biomarker prevalence without molecular confirmation of biomarker status, or any tumor type with molecular confirmation of biomarker status; For MTD cohort expansion, only dedifferentiated liposarcoma will be included.
* Presence of locally advanced or metastatic disease with at least one measurable lesion.

Exclusion criteria:

* Age <18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of >1.
* Life expectancy <12 weeks.
* Unstable brain or leptomeningeal disease based on history and physical examination.
* Inadequate organ functions, positive pregnancy test.
* Pregnancy or breast-feeding.
* Any anti-cancer drug therapy within 2 weeks (8 weeks for mitomycin C or nitrosoureas) or 5 half-lives of the drug prior to study treatment, whichever is shorter, prior to study treatment.
* Unwillingness, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ an effective barrier or medical method of contraception during the study drug administration and follow-up periods.
* Recent (3 months) history of acute pancreatitis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-07-13; Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
SAR405838 Maximum tolerated dose (MTD) | Cycle 1 (21 days) or 2 Cycles (42 days) dependent on dosing schedule
In MTD cohort, clinical benefit | Until disease progression

SECONDARY OUTCOMES:
Adverse events (eg, number of patients experiencing AEs) | Baseline to end of study
PK parameters (Cmax, Tmax, AUC) | Baseline to end of study
Biomarkers | Baseline to end of study
Clinical response | Baseline to end of study
Drug administration compliance | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States (3):
  - Investigational Site Number 840101, Boston, Massachusetts
  - Investigational Site Number 840001, Boston, Massachusetts
  - Investigational Site Number 840002, New York, New York
- Investigational Site Number 250001, Villejuif, France
- Netherlands (3):
  - Investigational Site Number 528001, Amsterdam
  - Investigational Site Number 528003, Rotterdam
  - Investigational Site Number 528002, Utrecht

REFERENCES:
- [Derived] de Jonge M, de Weger VA, Dickson MA, Langenberg M, Le Cesne A, Wagner AJ, Hsu K, Zheng W, Mace S, Tuffal G, Thomas K, Schellens JH. A phase I study of SAR405838, a novel human double minute 2 (HDM2) antagonist, in patients with solid tumours. Eur J Cancer. 2017 May;76:144-151. doi: 10.1016/j.ejca.2017.02.005. Epub 2017 Mar 17. PMID 28324749